CLINICAL TRIAL: NCT03617861
Title: Effect of Secretin on Gastric Accommodation, Emptying and Post-nutrient Challenge Symptoms in Functional Dyspepsia and Healthy Subjects
Brief Title: Effect of Secretin in Functional Dyspepsia and Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Professor and Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-003744; R01DK115950 (NIH); R01DK122280 (NIH); UL1TR002377 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Dyspepsia; Healthy
MeSH Terms: conditions — Dyspepsia | interventions — Secretin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Controls: Secretin Then Placebo (Experimental): Healthy subjects first receive human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the placebo treatment (normal saline, matching Secretin dose) via IV over 1 min on Visit Day 2.
  Interventions: Drug: Human Secretin; Drug: Placebo
- Healthy Controls: Placebo Then Secretin (Experimental): Healthy subjects first receive placebo treatment (normal saline, matching Secretin dose) via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 2.
  Interventions: Drug: Human Secretin; Drug: Placebo
- Functional Dyspepsia: Secretin Then Placebo (Experimental): Functional Dyspepsia subjects first receive human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the placebo treatment (normal saline, matching Secretin dose) via IV over 1 min on Visit Day 2.
  Interventions: Drug: Human Secretin; Drug: Placebo
- Functional Dyspepsia: Placebo Then Secretin (Experimental): Functional Dyspepsia subjects first receive placebo treatment (normal saline, matching Secretin dose) via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 2.
  Interventions: Drug: Human Secretin; Drug: Placebo

INTERVENTIONS:
Drug: Human Secretin — Injected once over one minute
  Other Names: ChiRhoStim
Drug: Placebo — Injected once over one minute
  Other Names: Normal Saline

SUMMARY:
Insights into the pathophysiology of functional dyspepsia, with recent demonstration of inflammation with eosinophilia and mastocytosis in the duodenum (3, 6, 7), providing a possible lead toward reduced secretion of a potential mediator of post-prandial gastric accommodation, the gastrointestinal peptide hormone secretin. The dominant site of synthesis and secretion of this hormone are enteroendocrine S cells in the duodenum. Inflammation-induced damage to these cells could produce a deficiency. Since intraluminal acid is a prominent stimulant of S cell secretion, the attempts to treat functional dyspepsia with anti-secretory medications could actually exacerbate a secretin deficiency syndrome. This raises the possibility of the therapeutic use of a secretin agonist or a positive allosteric modulator of the secretin receptor for patients with functional dyspepsia.

DETAILED DESCRIPTION:
The investigators will utilize single photon emission computed tomography (SPECT) methodology and gamma scintigraphy present in the GI laboratory of the outpatient Clinical Research Unit to study fasting gastric volumes and postprandial gastric accommodation responses and gastric emptying rates of a standardized meal in patients with functional dyspepsia and healthy subjects. Both groups will be studied twice, using crossover design, once with administration of secretin and once with placebo.

ELIGIBILITY:
Patients with FD and prior documentation of normal or accelerated gastric emptying and/or reduced gastric accommodation.

Inclusion criteria:

* Able to provide written informed consent prior to any study procedures and be willing and able to comply with study procedures
* No medical problems or chronic diseases, other than functional dyspepsia, for that group
* Body mass index of 18-35 kg/m2
* Female subjects must have negative urine pregnancy tests and must not be lactating prior to receiving study medication and radiation exposure. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female subjects unable to bear children must have this documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)].

Exclusion criteria:

* Unable or unwilling to provide informed consent or to comply with study procedures
* Diagnosis of other gastrointestinal diseases besides functional dyspepsia
* Structural or metabolic diseases that affect the GI system
* Unable to avoid the following over-the-counter medications 48 hours prior to the baseline period and throughout the study:

  * Medications that alter GI transit or motor function including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin, buspirone, clonidine, tricyclic antidepressants, and secretin-norepinephrine reuptake inhibitors
  * Analgesic drugs including NSAIDs and COX-2 inhibitors
  * NOTE: Stable doses of thyroid replacement, estrogen replacement, low-dose aspirin for cardio-protection, low stable dose antidepressants of the SSRI class, and birth control (but with adequate backup contraception, as drug interactions with birth control have not been conducted) are permissible.
* History of recent surgery (within 60 days of screening)
* Acute or chronic illness or history of illness which in the opinion of the investigator could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data, such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
* Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the investigator
* Acute GI illness within 48 hours of initiation of the baseline period
* Females who are pregnant or breastfeeding
* History of excessive alcohol use or substance abuse
* Participation in an investigational study within the 30 days prior to dosing in the present study
* Any other reason, which in the opinion of the investigator, would confound proper interpretation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Brandler J, Miller LJ, Wang XJ, Burton D, Busciglio I, Arndt K, Harmsen WS, Camilleri M. Secretin effects on gastric functions, hormones and symptoms in functional dyspepsia and health: randomized crossover trial. Am J Physiol Gastrointest Liver Physiol. 2020 Apr 1;318(4):G635-G645. doi: 10.1152/ajpgi.00371.2019. Epub 2020 Feb 10. PMID 32036693
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Secretin Then Placebo: Healthy subjects first receive human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the placebo treatment (normal saline matching Secretin dose) via IV over 1 min on Visit Day 2.
- Healthy Controls: Placebo Then Secretin: Healthy subjects first receive placebo treatment (normal saline matching Secretin dose) via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 2.
- Functional Dyspepsia: Secretin Then Placebo: Functional Dyspepsia subjects first receive human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the placebo treatment (normal saline matching Secretin dose) via IV over 1 min on Visit Day 2.
- Functional Dyspepsia: Placebo Then Secretin: Functional Dyspepsia subjects first receive placebo treatment (normal saline matching Secretin dose) via IV over 1 min on Visit Day 1. After a 1 to 4 week washout period, they received the human Secretin 0.2 mcg/kg via IV over 1 min on Visit Day 2.
Period: First Intervention (1 Day)
Arm/Group | Healthy Controls: Secretin Then Placebo | Healthy Controls: Placebo Then Secretin | Functional Dyspepsia: Secretin Then Placebo | Functional Dyspepsia: Placebo Then Secretin
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout (1 to 4 Weeks)
Arm/Group | Healthy Controls: Secretin Then Placebo | Healthy Controls: Placebo Then Secretin | Functional Dyspepsia: Secretin Then Placebo | Functional Dyspepsia: Placebo Then Secretin
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Healthy Controls: Secretin Then Placebo | Healthy Controls: Placebo Then Secretin | Functional Dyspepsia: Secretin Then Placebo | Functional Dyspepsia: Placebo Then Secretin
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: Healthy controls were randomly assigned to secretin or placebo allocation before treatment. After a 1 to 4 week washout period, they received the alternate treatment from that administered on Day 1.
- Functional Dyspepsia: Functional Dyspepsia subjects were randomly assigned to secretin or placebo allocation before treatment. After a 1 to 4 week washout period, they received the alternate treatment from that administered on Day 1.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Functional Dyspepsia | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45.0 [38.0 to 49.0] | 50.5 [42.0 to 55.0] | 47.0 [40.0 to 52.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Satiation
Description: Thirty (30) minutes after ingesting the meal of 300 mL radio-labeled Ensure drink, an additional Ensure drink was ingested at a constant rate of 30 mL/min until maximum tolerated volume was reached.
Time Frame: 60 minutes
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Healthy Controls: Secretin: Healthy controls who received human Secretin 0.2 mcg/kg via IV over 1 min on either the first or second study visit day.
- Healthy Controls: Placebo: Healthy controls who received placebo treatment (normal saline matching Secretin dose) via IV over 1 min on either the first or second study visit day.
- Functional Dyspepsia: Secretin: Functional Dyspepsia subjects who received human Secretin 0.2 mcg/kg via IV over 1 min on either the first or second study visit day.
- Functional Dyspepsia: Placebo: Functional Dyspepsia subjects who received placebo treatment (normal saline matching Secretin dose) via IV over 1 min on either the first or second study visit day.
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
mL | 892.5 [892.5 to 1011] | 951.75 [892.5 to 1129.5] | 655.5 [537 to 774] | 892.5 [655.5 to 1011]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.0574, ANCOVA

2. Primary Outcome: Fasting Gastric Volume
Description: Gastric fasting volume was measured prior to a meal of 300 mL standardized radio-labeled Ensure drink using an intravenous injection of Technetium Tc-99m pertechnetate and noninvasive single photon emission-computed tomography (SPECT).
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
mL | 171.28 [146.17 to 189.39] | 152.96 [145.5 to 161.04] | 227 [186.7 to 251.2] | 210.2 [179.38 to 240.54]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.1451, ANCOVA

3. Primary Outcome: Postprandial Volume
Description: Postprandial volume was measured 15 minutes after ingestion of 300 mL standardized radio-labeled Ensure drink using an intravenous injection of Technetium Tc-99m pertechnetate and noninvasive single photon emission-computed tomography (SPECT).
Time Frame: 15 minutes
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
mL | 435.85 [384.70 to 647.71] | 457.43 [329.39 to 495.01] | 593.80 [557.85 to 637.90] | 582.36 [546.51 to 631.33]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.85, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.4233, ANCOVA

4. Primary Outcome: Change in Gastric Accommodation
Description: The change in gastric accommodation was measured in mL using the difference between the fasting gastric volume and the postprandial volume.
Time Frame: Baseline, 30 minutes
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
mL | 270.44 [221.97 to 468.01] | 271.01 [194.74 to 343.62] | 378.6 [339.42 to 404.18] | 370.2 [339.09 to 382.06]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.92, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.3891, ANCOVA

5. Primary Outcome: Gastric Emptying
Description: Gastric emptying was measured via scintigraphy 30 minutes after ingestion of 300 mL of radio-labeled Ensure drink and was reported as the percentage of the radio-labeled liquid meal emptied from the stomach.
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: percentage of gastric emptying
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of gastric emptying | 7.0 [0 to 10.0] | 19.0 [15.0 to 26.0] | 0 [0 to 0] | 8.0 [2.0 to 9.0]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Healthy Secretin vs Healthy Placebo; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Healthy vs Functional Dyspepsia; Test type: Superiority; p = 0.0355, ANCOVA

6. Primary Outcome: Change in Postprandial Symptoms
Description: 30 minutes after ingesting a meal of 300 mL of Ensure drink postprandial symptoms of fullness, nausea, bloating and pain were measured using a horizontal visual analog scales from 0 to 100, where 0 was 'none' and 100 was 'worst ever'.
Time Frame: Baseline, 30 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale
  Nausea | 1.5 [0 to 3] | 1.5 [0 to 2] | 10 [8 to 28] | 4 [4 to 11]
  Fullness | 7 [3 to 10] | 4.5 [2 to 6] | 31 [22 to 42] | 11 [5 to 33]
  Bloating | 1.5 [0 to 7] | 1.5 [0 to 3] | 24 [6 to 34] | 26 [8 to 28]
  Abdominal pain | 1 [0 to 2] | 2 [0 to 3] | 5 [2 to 19] | 10 [5 to 21]
Statistical Analysis 1: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Nausea: Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Nausea: Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Nausea: Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.0016, ANCOVA
Statistical Analysis 4: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Fullness: Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Fullness: Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.30, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Fullness: Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.0002, ANCOVA
Statistical Analysis 7: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Bloating: Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.41, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Bloating Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Bloating: Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.0330, ANCOVA
Statistical Analysis 10: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo; Abdominal Pain: Healthy Controls Secretin vs Healthy Controls Placebo; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Abdominal Pain: Functional Dyspepsia Secretin vs Functional Dyspepsia Placebo; Test type: Superiority; p = 0.57, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Healthy Controls: Secretin vs Healthy Controls: Placebo vs Functional Dyspepsia: Secretin vs Functional Dyspepsia: Placebo; Abdominal Pain: Healthy Controls vs Functional Dyspepsia; Test type: Superiority; p = 0.2375, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events will be collected on each patient for each of the two individual study days, over a total duration of approximately one year.
Groups:
- Healthy Controls: Secretin: Healthy controls who received human Secretin 0.2 mcg/kg via IV over 1 min.
- Healthy Controls: Placebo: Healthy controls who received placebo treatment (normal saline matching Secretin dose) via IV over 1 min.
- Functional Dyspepsia: Secretin: Functional Dyspepsia subjects who received human Secretin 0.2 mcg/kg via IV over 1 min.
- Functional Dyspepsia: Placebo: Functional Dyspepsia subjects who received placebo treatment (normal saline matching Secretin dose) via IV over 1 min.
Arm/Group | Healthy Controls: Secretin | Healthy Controls: Placebo | Functional Dyspepsia: Secretin | Functional Dyspepsia: Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls: Secretin (N=10) | Healthy Controls: Placebo (N=10) | Functional Dyspepsia: Secretin (N=10) | Functional Dyspepsia: Placebo (N=10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Postprandial fullness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT03617861/Prot_SAP_000.pdf